CLINICAL TRIAL: NCT02713919
Title: Mixed Methods Study to Test the Efficacy of the Adapted German PRO-SELF® Plus Pain Control Program, an Intervention Directed at Outpatients With Cancer and Their Family Caregivers to Reduce Pain and Related Symptoms
Brief Title: Study to Test the Efficacy of the PRO-SELF® Plus Pain Control Program to Reduce Pain in Outpatients With Cancer
Acronym: PEINCA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient enrollment rate
Sponsor: Elisabeth Spichiger (Other)
Collaborators: University Hospital, Zürich (Other); Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Elisabeth Spichiger, Lecturer, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Multicenter PEINCA
Record Dates: First submitted 2016-03-08; First posted 2016-03-21 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Pain Management
Keywords: Cancer; Outpatients; Family Caregivers
MeSH Terms: conditions — Agnosia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Adapted German PRO-SELF© Plus Pain Control Program
  Interventions: Behavioral: Adapted German PRO-SELF© Plus Pain Control Program
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Adapted German PRO-SELF© Plus Pain Control Program — Two in-home visits (60 minutes) with at least weekly follow-up (visit or telephone call according to algorithm): Structured and tailored components; review of pain diary with participant, provision of information on pain medication, nurse coaching regarding pain self-management, detailed side-effect management plan, if distressing side-effects arise, re-evaluation together with participant at each subsequent visit.
  Arms: Intervention Group

SUMMARY:
Background: Up to 64% of cancer patients experience pain, and as many as 40% of patients with pain do not receive adequate pain management. And while potential to reduce pain has been shown in several interventions that support patients' self-management, effects have been moderate. Purpose: This multicenter mixed methods study primarily aims to evaluate the efficacy of the adapted German PRO-SELF© Plus Pain Control Program (PCP) on pain intensity, to explore the intervention's effect on associated symptoms and other patient and family caregiver (FC) outcomes, and to explore patients' and FCs' experiences with cancer pain management.

Methods: A nested concurrent mixed methods design will be used for this multi-center study, that is, a randomized controlled trial (RCT) will be combined with a qualitative substudy. Participants will be randomly assigned to a 6-week intervention or usual care group; outcomes will be evaluated at 6 weeks post-randomization. The primary outcome will be pain intensity. A total sample of 210 patients with cancer pain and approximately 105 FCs will be recruited from the oncology outpatient clinics of the University Hospitals Basel, Zurich and Bern. The intervention is designed to implement structured and tailored components (information, skill-building, nurse coaching) and aims at improving patients' pain self-management. Data analysis will follow an intent-to-treat strategy and generalized mixed models will be used. For the qualitative substudy, 60 patients and FCs of both groups will be interviewed. Data will be systematically summarized.

DETAILED DESCRIPTION:
Background: Between 33% and 64% of cancer patients experience pain; however, despite effective treatment options, as many as 40% of patients with pain do not receive adequate pain management. And while potential to reduce pain has been shown in several interventions that support patients' self-management of cancer pain, effects to date have been moderate. However, in a recent randomized controlled trial (RCT), Miaskowski's PRO-SELF© Pain Control Program (PCP) showed statistically and clinically significant pain reduction. This intervention was subsequently adapted for a second trial as PRO SELF© Plus PCP. The planned multi-center mixed methods study is based on this earlier work. In our previous pilot study, the PRO-SELF© Plus PCP was translated and adapted for a German speaking population. The feasibility of the intervention and study procedures was established and the intervention enhanced based on the pilot study's implications.

Purpose: This multi-center mixed methods study aims (1) to evaluate the efficacy of the adapted German PRO-SELF© Plus PCP, designed to improve outpatients' and their family caregivers' (FCs) management of pain on pain intensity; (2) to explore the intervention's effect on associated symptoms and other patient and FC outcomes; (3) to explore patients' and FCs' experiences with cancer pain management in both the intervention group and the usual care group; and (4) to interpret quantitative and qualitative findings and eventually synthesize them. To our knowledge, this will be the first evaluation of an intervention to support pain self-management in German speaking outpatients with cancer related pain and their FCs.

Methods: A nested concurrent mixed methods design will be used for this multi-center study, that is, an RCT will be combined with a qualitative substudy. Participants will complete a baseline evaluation, after which they will be randomly assigned to a 6-week intervention or usual care group. Blinding of data collectors is not feasible. Participants in both groups will complete a daily pain and symptom diary; other outcomes will be evaluated at 6 weeks post-randomization. The primary outcome of this study will be average and worst pain intensity. A total sample of 210 patients with cancer pain and approximately 105 FCs will be recruited from the oncology outpatient clinics of the University Hospitals Basel, Zurich and Bern. The intervention is designed to implement structured and tailored components (information, skill-building, nurse coaching) of the German PRO-SELF© Plus PCP. Participants will receive weekly in-home or telephone visits. Data analysis will follow an intent-to-treat strategy and generalized mixed models will be used. Average per-patient costs for the intervention will be calculated. For the qualitative substudy, approximately 7-10 patients and FCs per group and site will be interviewed regarding their experiences with pain management and intervention. Interpretive description will be used, including stepwise, systematic and iterative processing of data, leading to a meaningful description and interpretation.

Significance: The planned RCT will test the efficacy of the adapted German PRO-SELF© Plus PCP, with findings from the qualitative substudy providing additional insights. Qualitative results will support the interpretation of quantitative results and vice versa. If efficacious in decreasing average and worst pain in patients with cancer by improving patients' and FCs' pain self-management, the adapted German PRO-SELF© Plus PCP could be adapted to and implemented in clinical practice. Specially trained oncology nurses in outpatient clinics and home care organizations could apply the intervention as needed.

ELIGIBILITY:
Patient Inclusion Criteria:

* any type of cancer pain, including bone metastasis, somatic or visceral pain, with repeated pain ≥ 3 on a 0-10 Numeric Rating Scale (NRS) during the last week
* estimated life expectancy of > 6 months as assessed by the physician
* 18 years of age or older
* being able to understand, read and write German
* access to a telephone
* living within one hour's driving distance of a participating site

Adapted inclusion criterion (from 01 Sept 2016 on)

- any type of cancer pain, including bone metastasis, somatic or visceral pain, with repeated pain ≥ 3 on a 0-10 Numeric Rating Scale (NRS) during the last week

Patient Exclusion Criteria:

* cognitive dysfunction (as assessed by the physician) that would preclude full participation
* hearing impairment that precludes telephone conversations
* solely neuropathic pain (as assessed by the physician)
* participation in another clinical trial that requires extended hospitalizations (> 2 weeks)
* participation in another clinical trial that could exert an influence on the study intervention's effectiveness
* Family caregiver (FC) involved in pain management who declines to participate in the intervention (FCs are not required to participate in the study as participants).

FC Inclusion Criteria:

* 18 years of age or older
* being able to understand, speak and write German; and
* willingness to participate in all intervention sessions

FC Exclusion Criterion:

* hearing impairment that precludes understanding telephone conversation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-04-22 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Change in average and worst pain intensity | daily during weeks 0 - 6
  Measurement of Change in pain intensity using a numeric rating scale, 0-10,with 0 = no pain, 10 = worst imaginable pain

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Spichiger, PhD, Principal Investigator — University Basel, Medical Faculty, Institute of Nursing Science; Horst Rettke, PhD, Study Director — University Hospital Zurich, Center Clinical Nursing Science
Locations (3):
- Switzerland (3):
  - University Hospital Basel, Basel
  - Inselspital Bern University Hospital, Bern
  - University Hospital Zurich, Zurich

REFERENCES:
- [Derived] Valenta S, Miaskowski C, Spirig R, Zaugg K, Denhaerynck K, Rettke H, Spichiger E. Randomized clinical trial to evaluate a cancer pain self-management intervention for outpatients. Asia Pac J Oncol Nurs. 2022 Jan 21;9(1):39-47. doi: 10.1016/j.apjon.2021.12.003. eCollection 2022 Jan. PMID 35528799
- [Derived] Valenta S, Spirig R, Miaskowski C, Zaugg K, Spichiger E. Testing a pain self-management intervention by exploring reduction of analgesics' side effects in cancer outpatients and the involvement of family caregivers: a study protocol (PEINCA-FAM). BMC Nurs. 2018 Dec 12;17:54. doi: 10.1186/s12912-018-0323-x. eCollection 2018. PMID 30559603